CLINICAL TRIAL: NCT07050173
Title: Patients With Repetitive Head Impact Orally Supplemented With Gamma-glutamylcysteine: An Open Label Trial With MR Spectroscopy and Neuropsychological Testing
Brief Title: Monitoring Patients With Repetitive Head Impact With Gamma-glutamylcysteine Supplementation
Acronym: RHIGSH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pravat Mandal (Other)
Collaborators: Chuck Noll Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Pravat Mandal, Research Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY24120016; 0025 (Other: Chuck Noll Foundation)
Record Dates: First submitted 2025-06-20; First posted 2025-07-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Repetitive Head Impacts
Keywords: Brain injury; Glutathione; MR spectroscopy; Non- invasive; GGC; RHI; TES; Brain; Blood
MeSH Terms: conditions — Brain Injuries | interventions — gamma-glutamylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gamma - Glutamylcystiene (Experimental): Each participant will receive gamma-glutamyl cysteine (GGC) tablet orally 400mg (two times) per day once in the morning and once in the evening for 12 months.
  Interventions: Drug: Gamma-glutamylcysteine (GGC)

INTERVENTIONS:
Drug: Gamma-glutamylcysteine (GGC) — 400mg tablet orally (two times) per day.
  Other Names: GGC

SUMMARY:
The goal of this clinical trial is to test whether the gamma - glutamylcystiene (GGC) oral supplement can reach the brain and subsequently increase antioxidant glutathione (GSH) level in people with repetitive head impact (RHI). This will reduce the oxidative stress related injury in people with RHI.This unique study's main objective is to test the:

1. Change in GSH in brain and blood levels through GGC supplementation.
2. Change in the cognitive function in RHI patients due to GGC supplementation.

DETAILED DESCRIPTION:
This study is designed to evaluate the effects of GGC supplementation in patients with a history of repetitive head impacts (RHI) who are at risk for developing Traumatic Encephalopathy Syndrome (TES). The trial will include specific individuals who satisfy the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Retired NFL player, retired Navy SEAL/army personnel with combat experience exposed to repetitive head impact;
* Memory and behavioral complaint per self- or informant-report;
* Age (30 to 70 years of age) years;
* Able to read and write in English and to give consent to participate in the study.

Exclusion Criteria:

* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments in the eyes, skin, or body.
* Subjects with claustrophobia.
* Subject with mild cognitive impairment [TICS score of 29 or lower OR >=1.0 standard deviations below age-expectation on at least two cognitive members within the same cognitive domain (e.g. memory, attention, etc.) on the baseline neuropsychological testing;
* Subjects with a history of cancer;
* Subjects with active psychosis or delirium;
* Subjects with chronic kidney (creatinine > 1.5mg/dL) or liver disease (AST ≥ 1.5 ULN; ALT ≥1.5 ULN) within 30 days prior to enrollment;
* Subjects on antioxidant therapy (gingko biloba or N-acetylcysteine) or illicit drug abuse/dependence (cocaine, heroin, marijuana, or fentanyl;
* Repeated head injury patients with neurosurgical intervention and;
* Subjects with repeated head injury within the last 90 days.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
Changes in brain glutathione levels (mM) in people with Repetitive Head Injury (RHI) using Magnetic Resonance Spectroscopy in pre and post supplementation. | 12 months
  (MRS) is a non-invasive imaging technique, to detect various neurochemical (e.g. glutathione) using MEGA-PRESS sequence from 1H MR spectroscopy.
Changes in baseline blood glutathione levels (µmol/l) in people with RHI due to GGC supplementation. | 12 months
Changes in blood iron levels(ng/μl) in people with RHI due to GGC supplementation. | 12 months

SECONDARY OUTCOMES:
Correlation between glutathione and iron levels in the brain and blood with dysbiotic features of the gut microbiome in people with RHI. | 12 months
  Brain imaging, blood and stool samples will be collected to determine the correlation between glutathione and iron levels in the brain and blood with dysbiotic features of the gut microbiome in people with RHI.
Changes from baseline in the cognitive functions (immediate memory, visuospatial memory, language etc) using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) in people with RHI . | 12 months
  Interpretation: Higher scores > 70 indicate greater cognitive function (PMID =36648917)
Changes in brain iron levels (ppb) in people with RHI using susceptibility mapping between pre and post supplementation. | 12 months
Changes from baseline in the cognitive functions ( executive functions like attention, speed, and mental flexibility ) using Trail Making Test (TMT) A&B in people with RHI. | 12 months
  Scoring Method: The average scores are as follows:
  * Trail A - 29 seconds
  * Trail B - 75 seconds Interpretation: Higher scores indicate greater impairment
Changes from baseline in the cognitive functions and emotional well-being using Delis-Kaplan Executive Functioning System (D-KEFS) Color Word Interference test in people with a RHI | 12 months
  Interpretation: Higher score (> 7) (PMID=21122190) indicates greater executive functions which includes cognitive abilities essential for tasks such as planning, problem-solving, and decision-making.
Changes from baseline in the cognitive functions and emotional well-being using Test of Premorbid Functioning (TOPF ) in people with RHI (PMID=36648917) | 12 months
  Interpretation of the results: Higher scores (>45 above 315191110 indicate better cognitive and memory function.
Changes from baseline in the cognitive functions and emotional wellbeing using Brief Symptom Inventory (BSI-18) (self-report) in people RHI . | 12 months
  Scoring Method: Each item is scored on a 0-4 scale, with the total score indicating the severity of distress.
  Interpretation: Higher total scores indicate greater severity of psychological distress.
Changes from baseline in the cognitive functions and emotional well-being using PROMIS Cognitive Function -Short Form 8a (self-report) tool in people RHI. | 12 months
  Scoring Method:
  Raw Score: 8-40 Interpretation: Lower scores on this measure indicate greater subjective cognitive difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Pravat K Mandal, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical study report data will be provided after the study data is analyzed and published. A comprehensive report will be sent to the IRB. The respective agency will be reported accordingly. Requests for the release of data must be submitted in writing to the PI, clearly stating the purpose of the request, the specific data needed, and the intended use. The PI, in collaboration with the research team, will review each request to ensure compliance with institutional policies, ethical standards, and any relevant data use agreements.
Supporting Information: CSR

REFERENCES:
- [Background] Mandal PK, Dwivedi D, Joon S, Goel A, Ahasan Z, Maroon JC, Singh P, Saxena R, Roy RG. Quantitation of Brain and Blood Glutathione and Iron in Healthy Age Groups Using Biophysical and In Vivo MR Spectroscopy: Potential Clinical Application. ACS Chem Neurosci. 2023 Jun 21;14(12):2375-2384. doi: 10.1021/acschemneuro.3c00168. Epub 2023 May 31. PMID 37257017
- [Background] Mandal PK, Saharan S, Tripathi M, Murari G. Brain glutathione levels--a novel biomarker for mild cognitive impairment and Alzheimer's disease. Biol Psychiatry. 2015 Nov 15;78(10):702-10. doi: 10.1016/j.biopsych.2015.04.005. Epub 2015 Apr 14. PMID 26003861